CLINICAL TRIAL: NCT03965546
Title: Clinical Study of ET 140202 -T Cell Combined With TAE or Sorafenib in the Treatment of Advanced Liver Cancer
Brief Title: ET 140202 -T Cell Combined With TAE or Sorafenib in the Treatment of Liver Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Eureka Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019（ZD13）
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-05

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer; Liver Neoplasms; Metastatic Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ET140202-T cell combine with Sorafenib (Experimental): Sorafenib treatment everyday and autologous ET140202-T cell administered by intravenous (IV) infusion
  Interventions: Combination Product: Sorafenib combined with ET140202-T cell
- ET140202-T cell combine with TAE (Experimental): TAE treatment ahead every two times of autologous ET140202-T cell administered by intravenous (IV) infusion
  Interventions: Combination Product: TAE combined with ET140202-T cell
- solo ET140202-T cell (Experimental): autologous ET140202-T cell administered by intravenous (IV) infusion
  Interventions: Biological: ET140202-T cell

INTERVENTIONS:
Combination Product: Sorafenib combined with ET140202-T cell — 1. Sorafenib starting dose of 400mg b.i.d. a.c.
  2. Autologous T cells transduced with lentivirus encoding an anti-AFP (ET140202) expression construct by intravenous (IV) infusion
  Arms: ET140202-T cell combine with Sorafenib
Combination Product: TAE combined with ET140202-T cell — 1. Transarterial embolization(TAE) treatment
  2. Autologous T cells transduced with lentivirus encoding an anti-AFP (ET140202) expression construct -intravenous (i.v.)
  Arms: ET140202-T cell combine with TAE
Biological: ET140202-T cell — Autologous T cells transduced with lentivirus encoding an anti-AFP (ET140202) - expression construct -intravenous (i.v.)
  Arms: solo ET140202-T cell

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ET 140202 -T cell combined With TAE or Sorafenib in the treatment of liver cancer

DETAILED DESCRIPTION:
The molecular target for ET140202-T cells is HLA-A02 complexed with a HLA-A02-restricted peptide of alpha fetoprotein (AFP), which is expressed on 60-80 percent of hepatocellular carcinoma (HCC). This clinical study evaluates the safety and pharmacokinetics of ET140202-T cells with TAE or Sorafenib in patients with HCC who have no available curative therapeutic options and a poor overall prognosis.

ELIGIBILITY:
Inclusion Criteria:

* AFP-expressing HCC and serum AFP >10 x ULN
* Abandon or failure in first or second line treatment
* Molecular HLA class I typing confirms participant carries at least one HLA-A02 allele
* Child-Pugh score of A or B, ECOG 0-2, Life expectancy > 6 months
* Measurable disease as defined by: at least 1 liver lesion that can be accurately and serially measured.
* Negative serum pregnancy test for women with childbearing potential
* Adequate organ function as defined below:

  1. A pretreatment measured creatinine clearance (absolute value) of ≥50 ml/minute.
  2. Patients must have a serum direct bilirubin ≤3 x ULN, ALT and AST ≤5 x ULN.
  3. Ejection Fraction measured by echocardiogram or MUGA >50% (evaluation done within 6 weeks of screening does not need to be repeated)
  4. DLCO or FEV1 >45% predicted
  5. Absolute neutrophil count (ANC) ≥ 1500/mm3 (10^9/L), Platelet count ≥ 50,000/mm3 (10^9/L)
  6. INR ≤1.5 x ULN
  7. Informed Consent/Assent: All subjects must have the ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Patients with decompensated cirrhosis: Child-Pugh Score C
* Patients with tumor infiltration in the portal vein, hepatic veins or inferior vena cava that completely blocks circulation in liver.
* Patients with an organ transplantation history
* Patients with dependence on corticosteroids
* Patients with active autoimmune diseases requiring systemic immunosuppressive therapy
* Patients who are currently receiving or received within past 30 days anti-cancer therapy, local treatments for liver tumors (radiotherapy, embolism, ablation) or liver surgery
* Patients currently receiving other investigational treatments (biotherapy, chemotherapy, or radiotherapy)
* Participants with other active malignancies (except non-melanoma skin cancer and cervical cancer) within two years. Patients with a history of successfully-treated tumors with no sign of recurrence in the last two years may be enrolled.
* Patients with other uncontrolled diseases, such as active infections Acute or chronic active hepatitis B or hepatitis C.
* Women who are pregnant or breast-feed
* HIV-infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2019-05-30 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Frequency of ARTEMIS T cell treatment-related adverse events | 28 days up to 2 years
  Include but not limited to: Fever, chills, nausea, vomiting, jaundice and other gastrointestinal symptoms; Fatigue, hypotension, respiratory distress; Tumor lysis syndrome; Cytokine release syndrome; Neutropenia, thrombocytopenia; Liver and kidney dysfunction. Assessed at all visits.

SECONDARY OUTCOMES:
Rate of disease response by RECIST in the liver | 2 years
  Response rates will be estimated as the percent of patients with objective response (OR)，which was defined as any of complete remission (CR), partial response (PR) at 2 years.
Rate of disease response by RECIST at non-liver sites | 2 years
  Response rates will be estimated as the percent of patients with objective response (OR), complete remission (CR), partial response (PR), stable disease (SD), no response (NR), overall survival (OS).
Progression free survival (PFS) | at 4 months, 1 year, 2 years
  Progression free survival (PFS) at 4 months, 1 year and 2 years
Median Survival（MS） | at 4 months, 1 year, 2 years
  Median Survival（MS）at 4 months, 1 year and 2 years
Overall survival（OS） | at 2 years
  overall survival（OS）at 2 years
AFP serum levels | 2 years
  Percent change compared to the baseline
Number of ET140202-T cells in peripheral blood | 2 years
  Number of ET140202-T cells in peripheral blood will be presented as Time to peak, Time to baseline level
Alpha-fetoprotein (AFP) expression in tumors | 4-8 weeks
  Percent of AFP-positive cells in randomly selected fields in tumor biopsies.
IL-6 serum levels | 4-8 weeks
  Amount change compared to the baseline
IL-2 serum levels | 4-8 weeks
  Amount change compared to the baseline
IL-10 serum levels | 4-8 weeks
  Amount change compared to the baseline
TNF-α serum levels | 4-8 weeks
  Amount change compared to the baseline
IFN-γ serum levels | 4-8 weeks
  Amount change compared to the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Xue Hui, PHD, Study Chair — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided